CLINICAL TRIAL: NCT06868368
Title: Perceptions of Vaping Products Among Young Adults
Brief Title: Perceptions of Vaping Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Alayna Tackett, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: OSU-24276; NCI-2024-10267 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2025-01-14; First posted 2025-03-10 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-09

CONDITIONS: Abuse Tobacco; Exposure
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Intervention Model Description: Randomization to condition order will be completed prior to study Visit 1. Each participant will receive a randomized ordering developed using a random sequence generator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Participant's personal nicotine e-cigarette (Active Comparator): The study participant's own preferred e-cigarette will be used for this condition.
  Interventions: Other: Biospecimen Collection; Other: Survey Administration; Behavioral: Vaping Topography; Other: Participant's Own Preferred E-cigarette
- Nicotine e-cigarette (Active Comparator): A fruit flavored commercially available nicotine e-cigarette will be used for this condition.
  Interventions: Other: Biospecimen Collection; Other: Survey Administration; Behavioral: Vaping Topography; Other: Nicotine E-cigarette
- 6-methyl nicotine (metatine) e-cigarette (Active Comparator): A fruit flavored commercially available metatine e-cigarette will be used for this condition.
  Interventions: Other: Biospecimen Collection; Other: Survey Administration; Behavioral: Vaping Topography; Other: 6-methyl-nicotine (metatine) e-cigarette

INTERVENTIONS:
Other: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection
Other: Survey Administration — Complete Surveys
Behavioral: Vaping Topography — Use e-cigarette connected to a topography device
Other: Participant's Own Preferred E-cigarette — Participant vapes their own preferred e-cigarette for 30 minutes
  Arms: Participant's personal nicotine e-cigarette
Other: Nicotine E-cigarette — Participant vapes a commercially available nicotine e-cigarette for 30 minutes
  Arms: Nicotine e-cigarette
Other: 6-methyl-nicotine (metatine) e-cigarette — Participant vapes a commercially available metatine e-cigarette for 30 minutes
  Arms: 6-methyl nicotine (metatine) e-cigarette

SUMMARY:
This clinical trial studies the effects, appeal, and abuse liability of 6-methyl nicotine (metatine) electronic cigarettes among young adults.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the pharmacokinetics of metatine and nicotine electronic (e)-cigarettes.

II. Assess the abuse liability and appeal of commercial e-cigarettes containing metatine versus nicotine.

III. Determine the impact of metatine on e-cigarette puffing behavior (topography).

OUTLINE: Participants attend 3 sessions where they will be randomized to 1 of 3 types of e-cigarette. Participants will use the e-cigarette ad-libitum for 30 minutes and answer survey questions about their perceptions of the e-cigarette. Participants must also undergo 4 blood draws during the vaping session.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21-34 years
* Current nicotine EC user (defined as ≥ weekly use over the past 3 months)
* Willing to provide informed consent and abstain from using any e-cigarette at least 12 hours prior to the three lab sessions
* Read and speak English

Exclusion Criteria:

* Recently coronavirus disease 2019 (COVID-19) positive (defined as a positive test in the past 30 days) or a recent COVID-19 hospitalization (defined as a hospitalization within the past 6 months)
* Unstable or significant psychiatric conditions (past and stable conditions will be allowed)
* History of cardiac event or distress within the past 3 months
* Have suffered from any serious lung disease or infection (e.g., tuberculosis, cystic fibrosis, or lung cancer) in the past 30 days
* Are currently pregnant, planning to become pregnant, or breastfeeding (will be verified with urine pregnancy test)
* Have hemophilia or another type of bleeding disorder
* Are blind, severely visually impaired, deaf, hard of hearing, or have a severe motor disability

Ages: 21 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-11-04 (Actual); Study Completion 2025-11-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of metatine and nicotine e-cigarettes | Pre-vaping session, Minute 5 of vaping session, Minute 15 of vaping session, Minute 30 of vaping session
  Pharmacokinetics of metatine and nicotine e-cigarettes will be examined by measuring the concentration of metatine and nicotine in blood plasma at different timepoints throughout the study vaping session.
E-cigarette puffing behavior | Week 1, Week 2, Week 3
  E-cigarette puffing behavior will be measured with a topography device that records frequency, duration, and flow rate of e-cigarette puffs. These measures are combined to inform the overall measure of e-cigarette puffing behavior.
Sensory perceptions of EC vaping experience | Minute 5 of vaping session, Minute 30 of vaping session
  Sensory perceptions of vaping will be measured by the Sensory E-cigarette Expectancies Scale (SEES) questionnaire. The SEES asks questions about sensory experiences associated with vaping on a scale from 0 (Never) - 4 (Almost Always).
Appeal ratings | Minute 5 of vaping session, Minute 30 of vaping session
  Participants will rate appeal (e.g., liking, disliking) on Visual Analogue Scales (range, 0-100).
Sensory ratings | Minute 5 of vaping session, Minute 30 of vaping session
  Participants will rate sensory attributes (e.g., harshness, coolness) on Visual Analogue Scales (range, 0-100).
Relief of withdrawal symptoms | Pre-vaping session, Minute 5 of Vaping Session, Minute 30 of vaping session
  Nicotine withdrawal relief will be measured by the Minnesota Nicotine Withdraw Scale (MNWS). The MNWS asks users how much they are currently feeling certain nicotine withdraw symptoms on a scale of None, Slight, Moderate, Mild, or Severe.

CONTACTS AND LOCATIONS:
Overall Officials: Alayna P Tackett, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu